CLINICAL TRIAL: NCT05564091
Title: Cataract Surgery in Conjunction With Ab-interno Canaloplasty Compared to Cataract Surgery Only in Patients With Mild to Moderate Primary Open-Angle Glaucoma
Acronym: CATALYST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Eye, Inc. (Industry)
Collaborators: Nova Eye Medical GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: NE 03021
Record Dates: First submitted 2022-09-29; First posted 2022-10-03 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Primary Open Angle Glaucoma
Keywords: Canaloplasty
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Cataract Extraction; Phacoemulsification

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Cataract surgery combined with ab-interno canaloplasty (Active Comparator): Ab-interno canaloplasty utilizing the iTrack Advance canaloplasty device (Nova Eye, Inc.)
  Interventions: Device: Cataract surgery combined with ab-interno canaloplasty utililzing the iTrack Advance canaloplasty device
- Control: Cataract surgery (Other): Cataract surgery alone
  Interventions: Procedure: Cataract surgery

INTERVENTIONS:
Device: Cataract surgery combined with ab-interno canaloplasty utililzing the iTrack Advance canaloplasty device — 360 degree microcatheterization and viscodilation of Schlemm's canal
  Arms: Cataract surgery combined with ab-interno canaloplasty
Procedure: Cataract surgery — Cataract surgery alone
  Other Names: Phacoemulsification
  Arms: Control: Cataract surgery

SUMMARY:
A prospective, multicenter, randomized, single-masked, post-market clinical trial comparing cataract surgery in conjunction with ab-interno canaloplasty utilizing the iTrack Advance canaloplasty device (Nova Eye, Inc.) to cataract surgery only in patients with mild to moderate, primary open angle glaucoma. Subjects will be followed for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate, primary open angle glaucoma
* Characteristics consistent with mild to moderate glaucoma
* Use of 1 - 4 ocular hypotensive medications at the Screening exam and meets the IOP (intraocular pressure) criteria
* Visually significant cataract

Exclusion Criteria:

Any of the following prior treatments for glaucoma (study eye):

* Laser Trabeculoplasty
* Endocyclophotocoagulation (ECP) or Micropulse laser
* iStent or iStent Inject
* Hydrus Microstent
* Trabeculectomy or other bleb forming procedure including Xen, Express, and glaucoma drainage device/valve.
* Prior canaloplasty (ab-interno and ab-externo)
* Prior goniotomy, or trabeculotomy (ab-interno or ab-externo)
* Suprachoroidal stent (e.g., Cypass, iStent Supra, XEN, MINIject)
* Concurrent IOP-lowering procedure other than use of the iTrackTM Advance canaloplasty device at the time of surgery (e.g., ECP, CPC, etc.)
* Previous treatment with iTrack (Note: permitted if fellow eye only was treated)
* Acute angle closure, traumatic, congenital, malignant, uveitic or neovascular glaucoma

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-09-08 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Reduction in mean Intraocular Pressure (IOP) at 12 months compared to baseline | 12 months
  IOP will be measured at each study visit using Goldmann applanation tonometry
Reduction in number of glaucoma medications at 12 months compared to baseline | 12 months
  The number of glaucoma medications will be recorded at 12 months compared to baseline

SECONDARY OUTCOMES:
Reduction in mean Intraocular Pressure (IOP) at 24-months compared to baseline | 24 months
  IOP will be measured at each study visit using Goldmann applanation tonometry
Reduction in glaucoma medications at 24-months compared to baseline | 24 months
  The number of glaucoma medications will be recorded at 24-months compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Koerber, MD, Principal Investigator — Augencentrum Köln Ophthalmology
Locations (4):
- Berkeley Eye Center, Sugar Land, Texas, United States
- Germany (3):
  - University of Bonn Eye Clinic, Bonn
  - Augencentrum Köln Ophthalmology, Cologne
  - St. Johannes Hospital, Dortmund

IPD SHARING:
Plan to Share IPD: No